CLINICAL TRIAL: NCT00072969
Title: A Randomized Trial of Recombinant Humanized Anti-IL-2 Receptor Antibody (Daclizumab) Versus Antithymocyte Globulin (ATG) to Treat the Cytopenia of Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040026; 04-H-0026
Record Dates: First submitted 2003-11-12; First posted 2003-11-13 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-08

CONDITIONS: Myelodysplastic Syndromes
Keywords: Immunosuppression; Myelodysplastic Syndrome; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Daclizumab

INTERVENTIONS:
Drug: Daclizumab

SUMMARY:
This study will evaluate a new immunosupressive therapy, Daclizumab, and compare it with antithymocyte globulin (ATG) to treat cytopenia, that is, the deficiency of cellular elements of the blood, in myelodysplastic syndrome (MDS). Daclizumab is an anti-interleukin-2 receptor (IL-2) antibody. MDS, also known as myelodysplasia, is a disorder that can cause anemia, spontaneous bleeding, and greater risk of infections. Although the bone marrow can still produce some blood cells, very few reach the bloodstream. The cause of MDS is not known, although its behavior is. Many patients need transfusions of red blood cells. They may also develop leukemia, which is often quite resistant to treatment with chemotherapy. However, the progression of the disorder to leukemia is usually slow, taking many years.

Patients 18 years of age and older who have MDS may be eligible for this study. Participants will undergo the following tests and procedures:

* Medical history and physical examination.
* Collection of blood for tests including blood counts, liver and kidney function, and antibodies against common viruses.
* Chest x-ray.
* Electrocardiogram.
* Bone marrow sample to confirm the diagnosis.

Participants will randomly receive either ATG or Daclizumab. If they are in the group to receive ATG, they will be admitted as inpatients to undergo the first 10 to 14 days of treatment. If they do not already have a catheter in one of the large veins of the neck, chest, or arm, one will be placed. ATG will be given through the catheter. Blood counts and other blood analysis will be monitored daily while the patients are treated. After about 10 days, they will be released, to be under the care of their referring physicians. Those participants who are in the group to receive Daclizumab will receive a total of five doses, one every 2 weeks, over 8 weeks, given through a vein as a 15-minute infusion. The first, third, and fifth dose will be given at the outpatient clinic. The second and fourth doses can be given either at the clinic or by the patients' primary hematologists.

All patients will be followed as outpatients at 3-month intervals for the first year, and then every 6 months for the next 3 years. Afterward, follow-up will be yearly. A small sample of blood will be drawn at the visits. Also, bone marrow examinations will be requested at the 6-month intervals for the first 3 years of treatment. If the treatment that patients are assigned to does not work, after 6 months, they will be eligible to receive the other treatment-provided that they have complied with the required blood tests and visits to the clinic required to assess the patients' safety.

DETAILED DESCRIPTION:
Many bone marrow failure syndromes in humans are now recognized to result from immunological mechanisms. These diseases include aplastic anemia, pure red cell aplasia, and some types of myelodysplasia. Patients with these conditions, who may suffer variable degrees of anemia, leukocytopenia, and thrombocytopenia, alone or in combination, have been shown to respond to a wide variety of immunosuppressive agents, ranging from corticosteroids to cyclosporine (CSA) and antithymocyte globulin (ATG), however, nonresponse and relapse continues to be a problem. Why some patients do not respond initially or others respond and then relapse is unclear. Autoreactive T cells may be resistant to the effect of ATG/CsA (nonresponders), while in others residual autoreactive T cells expand post-treatment leading to hematopoietic stem cell destruction and recurrent pancytopenia (relapse). Therefore, novel, less toxic immunosuppressive regimens that increase response rates and hematologic recovery and decrease relapse rates are needed.

One such novel therapy, Daclizumab, a humanized anti-interleukin-2 receptor (lL-2R) monoclonal antibody (mAb), acts against activated lymphocytes, thus sharing an important mechanism of action with ATG. The mAb is much less toxic than ATG and may be administered to outpatients at relatively infrequent intervals (every 2 weeks). Treatments with ATG alone and CsA alone have demonstrated varying degrees of success in alleviating the cytopenia of MDS. Our experience suggests that ATG rather than CSA is the more effective agent inducing hematological responses in susceptible MDS patients and that certain variables including the patient's age, whether or not they were HLA DR15, and days of red cell transfusion dependence prior to treatment were predictive of response.

We therefore propose this randomized phase II study to evaluate and compare a new immunosuppressive therapy, Daclizumab, with antithymocyte globulin (ATG) to treat the cytopenia of MDS in a population of subjects with intermediate or high predicted probability of response.

ELIGIBILITY:
INCLUSION CRITERIA:

MDS of RA, RARS & RAEB sub-types including those previously treated with chemotherapy or experimental agents such as retinoids, Vitamin D, and growth factors

Anemia requiring transfusion support with at least one unit of packed red blood cells per month for greater than or equal to 2 months

OR

thrombocytopenia (platelet count less than 50000/ul)

OR

neutropenia (absolute neutrophil count less than 500/ul).

Off all other treatments (except G-CSF, and transfusion support and related medications) for at least four weeks. G-CSF can be used before, during and after the protocol treatment for patients with documented neutropenia (less than 500/Ul) as long as they meet the criteria for anemia and/or thrombocytopenia as stated above.

ECOG performance status less than or equal to 2

High or intermediate predicted probability of response

EXCLUSION CRITERIA:

MDS of FAB sub-group chronic myelomonocytic leukemia (CMML)

Transformation to acute leukemia (FAB sub-group RAEB-T, ie, greater than 20% blasts in marrow aspirate)

Hypoplastic marrow without one major or two minor criteria

Treatment with growth factors (except for G-CSF) or cyclosporine within 4 weeks prior to entry to protocol

Recent or current treatment (24 hours wash out period) with the herbal supplement Echinacea purpurea or Usnea barbata (Old Man's Beard)

ECOG performance status of greater than 2

Active uncontrolled infection (chronic or current clinically significant infection, including hepatitis B or C virus infection)

Current pregnancy, or unwilling to take oral contraceptives or refrain from pregnancy if of childbearing potential

Patients for whom bone marrow transplant is indicated as standard therapy (age less than fifty-five with a fully-matched sibling donor)

Age less than 18 years

Not able to understand the investigational nature of the study or give informed consent

HIV positive patients

Active malignant disease (excluding basal cell carcinoma)

Serum creatinine greater than 2mg/dl

Patients who are moribund or patients with concurrent hepatic, renal, cardiac, metabolic, or any disease of such severity that death within 3 months is likely

Low predicted probability of response

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132
Dates: Start 2003-11; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Jonasova A, Neuwirtova R, Cermak J, Vozobulova V, Mocikova K, Siskova M, Hochova I. Cyclosporin A therapy in hypoplastic MDS patients and certain refractory anaemias without hypoplastic bone marrow. Br J Haematol. 1998 Feb;100(2):304-9. doi: 10.1046/j.1365-2141.1998.00551.x. PMID 9488617
- [Background] Biesma DH, van den Tweel JG, Verdonck LF. Immunosuppressive therapy for hypoplastic myelodysplastic syndrome. Cancer. 1997 Apr 15;79(8):1548-51. doi: 10.1002/(sici)1097-0142(19970415)79:83.0.co;2-y. PMID 9118037
- [Background] Nydegger UE. Suppressive and substitutive immunotherapy: an essay with a review of recent literature. Immunol Lett. 1985;9(4):185-90. doi: 10.1016/0165-2478(85)90031-8. No abstract available. PMID 3888832